CLINICAL TRIAL: NCT04714892
Title: Mechanisms Underlying Individual Variations of Taste and Smell in Obesity
Status: Recruiting | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000261; 000261-AA
Record Dates: First submitted 2021-01-16; First posted 2021-01-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08-07

CONDITIONS: Obesity
Keywords: chemosensation; Olfaction; Diet; obese; Perception; Natural History
MeSH Terms: conditions — Obesity; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: BMI of 18.5-29.9 kg/m2
- Obese: BMI of 30-39.9 kg/m2

SUMMARY:
Background:

Changes to the sense of taste or smell can change eating behavior. This may contribute to obesity. Researchers want to see how taste and smell perceptions that affect food choices may differ between people with obesity and without obesity.

Objective:

To understand the role that senses of taste and smell play in food intake.

Eligibility:

Adults ages 18-65 with obesity and without obesity

Design:

Participants will be screened with a medical history and physical exam. They will have a neurological and sensory exam. They will give blood and urine samples. They will be checked for previous SARS-CoV-2 infection. They will complete questionnaires about their eating habits, alcohol use, and smoking history.

Participants will have 2 study visits.

Participants will give stool, urine, blood, hair, nasal, and saliva samples. These samples will be used for gene testing.

Participants will have their weight, height, and hip and waist circumference measured. They will have an imaging scan that measures body composition.

Participants will complete questionnaires about their health, eating habits, and food preferences.

Participants will have taste tests and smell tests. They will have sensory tests to assess their response to stimuli.

Participants will have a dietary assessment. They will complete a food diary and a diet history questionnaire.

Participants will get a meal to eat. Data will be collected about their experience.

Participants will complete a sleep diary and wear a watch to measure their activity....

DETAILED DESCRIPTION:
Study Description:

This study involves comparison of taste and smell measures between obese and non-obese individuals. Taste and smell perceptions will be assessed in terms of their influence in food intake and food choices. We hypothesize that obesity negatively affects taste and smell perception thus affecting eating behavior.

Objectives:

Obesity is a major public health concern in America. An unhealthy diet is a recognized risk factor for the development of obesity. Public health efforts to modify eating behaviors have had limited success. Not only does an unhealthy diet contribute to obesity, but it can also lead to changes in gut microbiota that likely result in inflammation and changes in transcriptomic activity. Taste and smell perceptions, which can influence food choices and food consumption, may differ between obese and non-obese individuals. Currently, little is known about the underlying mechanisms causing variations in taste and smell systems in individuals with obesity, which limits the interventions currently available to address this critical issue. Findings from this study can be used to design more effective interventions for the prevention and treatment of obesity, to identify targets and strategies for countermeasures to prevent or improve obesity and its comorbidities, and to suggest ways to enhance dietary interventions. Moreover, findings will foster new lines of investigation for reducing risk of diet related conditions and for developing novel behavioral and pharmacological avenues of treatment and prevention. The proposed research is aligned with the overall mission of the National Institutes of Health to promote health and disease prevention. The findings from this study will ultimately lead to the development of personalized interventions for individuals with obesity and concurrent taste and smell alterations. Lastly, approaches included in this proposal are innovative and highly applicable to other complex health phenomena in which biological variations in inflammation and taste and smell perception impact an individual s health.

Endpoints:

Primary Endpoint: The primary dependent measures for this study are taste and olfaction measures.

Secondary Endpoints: Secondary measures include inflammatory markers, exosomes, microbiota, gene expression, DNA methylation, biological measures and personal factors.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Males and females between 18 to 65 years of age. Due to documented knowledge that taste and smell changes with age, we will limit the cohort within this age range.
* BMI between 18.5 and 29.9 kg/m^2 for healthy controls or between 30 and 39.9 kg/m^2 for obese subjects
* Fasted plasma glucose levels between 68-126 mg/dl or per Clinical Center ranges, and hemoglobin A1C<6.5%
* Able to provide his/her own consent
* Able to understand the protocol, as shown by scoring a 6 out of 6 on a consent quiz

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Because type-2 diabetic subjects have blunted taste responses, subjects with diagnosis of type II diabetes will be excluded.
* Hypoglycemic drug intake.
* Weight change of more than 15 pounds in the 6 months prior to screening
* Positive pregnancy test, currently pregnant or breastfeeding.
* Currently using any of the following medications: steroidal or nonsteroidal antiinflammatory medications, medications known to inhibit taste response (GLP1 agonists), antiepileptic or antidepressant agents, glucocorticoids, or antibiotics.
* Received a diagnosis by a medical professional of morbid obesity, liver or renal disease.
* Individuals with current heavy drinking. Women who drink 4 drinks or more in one occasion and 7 drinks in a week. Men who drink 5 drinks or more in one occasion and more than 14 drinks a week.
* Use of tobacco products or illicit drugs (as determined by urine drug screen and/or history/physical exam) in the last 30 days.
* Currently have an uncontrolled medical disorder (i.e., gastrointestinal, endocrine, cardiac, psychiatric).
* Any self-reported history of chronic rhinitis, eating disorder (including binge eating), chronic upper respiratory infection, chronic allergic rhinitis, or nasal polyps in the last 6 months of screening, or current daily use of nasal sprays.
* Abnormal complete blood count (CBC): White Blood Cell Count < 4 or > 10 K/uL, Red Blood Cell Count < 4 or > 7 M/uL, Hemoglobin < 12 g/dL for females or < 13 g/dL for males or any clinical signs/symptoms that indicate iron deficiency anemia per clinician s judgment at screening [National Heart, Lung and Blood Institute (NHLBI) definition (Anemia - Iron-Deficiency Anemia, Diagnosis NHLBI, NIH)].
* Bariatric surgery within the last 12 months of screening.
* History of cancer (e.g., head and neck cancer) and/or history of cancer treatment (e.g., radiotherapy to the head and neck area or chemotherapy).
* Altered cranial nerves identified by neurological evaluation during physical exam (screening visit).
* Currently experiencing temporary change/loss of taste and/or smell.
* Persistent loss of taste and/or smell due to COVID-19 or other reasons.
* Unable to read and understand English. Since all self-report measures are in English only, participants need to be able to read and understand the English language.
* NIAAA employees/staff or subordinates/relatives/co-workers of NIAAA employees/staff or study investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Washington DC metropolitan area and vicinity.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measures of taste and smell, and eating behavior | At enrollment
  Compare individuals with obesity to healthy controls in measures of taste and smell and eating behaviors.

SECONDARY OUTCOMES:
Inflammatory markers, exosome and microbiota | At enrollment
  Compare individuals with obesity to healthy controls in measures of inflammation (cytokines and chemokines) in circulating blood, and neuronally-derived exosomes from plasma, and in the oral and nasal microbiome composition and its metabolites.
Gene expression, DNA methylation, taste and smell measures | At enrollment
  Compare individuals with obesity to healthy controls on transcriptomic and epigenomic profiles in monocytes, based on gene expression (RNA sequencing) and whole genome DNA methylation, to identify associated variations in taste and smell perception.
Biological measures, personal factors, taste and smell measures | At enrollment
  Examine how biological measures of inflammation and genomic profiles relate to taste and smell variations based on personal factors (i.e., race, age, and sex) and other factors (i.e., diet) within the obese group
Severity of neuropsychological sysmptoms such as fatigue, anxiety, depression, sleep; perceived stress, pain and QoL | At enrollment
  Evaluate symptoms clusters with alterations in taste and smell and identify phenotypic symptoms characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Paule V Joseph, C.R.N.P., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share as stated in sharing plan of the protocol with proper MTAs in place.
Supporting Information: SAP, Analytic Code
Time Frame: Data may be available 5 years after the completion of the primary endpoint. Requests can be made by contacting the study PI.
Access Criteria: Data will be shared through restricted access to NIH-designated data repositories. Data and samples may be shared with investigators and institutions with an FWA or operating under the Declaration of Helsinki (DoH). Such sharing of data will be reported at the time of continuing review. Sharing with investigators without an FWA or not operating under the DoH will be submitted for prospective IRB approval. Submissions to NIH-sponsored or supported databases and repositories will be reported at the time of Continuing Review. Submission to non-NIH-sponsored or supported databases and repositories will be submitted for prospective IRB approval.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000261-AA.html